CLINICAL TRIAL: NCT04423211
Title: Phase III Study of Local or Systemic Therapy INtensification DIrected by PET in Prostate CAncer Patients With Post-ProstaTEctomy Biochemical Recurrence (INDICATE)
Brief Title: Treating Prostate Cancer That Has Come Back After Surgery With Apalutamide and Targeted Radiation Based on PET Imaging
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA8191; NCI-2020-02686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8191 (Other: ECOG-ACRIN Cancer Research Group); EA8191 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Conformal; apalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Congresses as Topic; Radiation; fluciclovine F-18; Goserelin; Radiotherapy, Intensity-Modulated; Leuprolide; luprolide acetate gel depot; Magnetic Resonance Spectroscopy; relugolix; Radiosurgery; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A (EBRT, short-term androgen deprivation therapy [STAD]) (Active Comparator): STEP 0: Patients undergo SOC PET/CT or PET/MR scan at baseline. Patients randomized to Arms C or D and receiving fluciclovine F18 IV undergo a repeat PET2 at time of PSA progression or clinical concerns for progression or 12 months after completion of enhanced systemic therapy, whichever occurs first. Patients in Arm C or D using another tracer for PET1 do not undergo PET2.
  STEP 1: Patients who are PET negative for extera pelvic metastases undergo SOC EBRT for 6 months. Patients also receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC for 6 months starting up to 3 months prior to EBRT but no later than 7 days after start of EBRT. All treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Computed Tomography; Drug: Degarelix; Radiation: External Beam Radiation Therapy; Other: Fluciclovine F18; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Relugolix; Drug: Triptorelin
- Arm B (EBRT, STAD, apalutamide) (Experimental): STEP 0: Patients undergo SOC PET/CT or PET/MR scan at baseline. Patients randomized to Arms C or D and receiving fluciclovine F18 IV undergo a repeat PET2 at time of PSA progression or clinical concerns for progression or 12 months after completion of enhanced systemic therapy, whichever occurs first. Patients in Arm C or D using another tracer for PET1 do not undergo PET2.
  STEP 1: Patients who are PET negative for extra pelvic metastases undergo SOC EBRT and receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC as in Arm A. Patients also receive apalutamide PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Apalutamide; Procedure: Computed Tomography; Drug: Degarelix; Radiation: External Beam Radiation Therapy; Other: Fluciclovine F18; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Relugolix; Drug: Triptorelin
- Arm C (EBRT, STAD, apalutamide) (Experimental): STEP 0: Patients undergo SOC PET/CT or PET/MR scan at baseline. Patients randomized to Arms C or D and receiving fluciclovine F18 IV undergo a repeat PET2 at time of PSA progression or clinical concerns for progression or 12 months after completion of enhanced systemic therapy, whichever occurs first. Patients in Arm C or D using another tracer for PET1 do not undergo PET2.
  STEP 1: Patients who are PET positive for extra pelvic metastases undergo SOC EBRT and receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC as in Arm A. Patients also receive apalutamide PO QD as in Arm B.
  Interventions: Drug: Apalutamide; Procedure: Computed Tomography; Drug: Degarelix; Radiation: External Beam Radiation Therapy; Other: Fluciclovine F18; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Relugolix; Drug: Triptorelin
- Arm D (EBRT, STAD, apalutamide, RT) (Experimental): STEP 0: Patients undergo SOC PET/CT or PET/MR scan at baseline. Patients randomized to Arms C or D and receiving fluciclovine F18 IV undergo a repeat PET2 at time of PSA progression or clinical concerns for progression or 12 months after completion of enhanced systemic therapy, whichever occurs first. Patients in Arm C or D using another tracer for PET1 do not undergo PET2.
  STEP 1: Patients who are PET positive for extra pelvic metastases undergo SOC EBRT and receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC as in Arm A and apalutamide PO QD as in Arm B. Patients also undergo SBRT or 3D CRT, IMRT (including VMAT), and IMPT over 3-10 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Apalutamide; Procedure: Computed Tomography; Drug: Degarelix; Radiation: External Beam Radiation Therapy; Other: Fluciclovine F18; Drug: Goserelin Acetate; Procedure: Intensity-Modulated Proton Therapy; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Relugolix; Radiation: Stereotactic Body Radiation Therapy; Drug: Triptorelin; Radiation: Volume Modulated Arc Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
  Arms: Arm D (EBRT, STAD, apalutamide, RT)
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
  Arms: Arm B (EBRT, STAD, apalutamide); Arm C (EBRT, STAD, apalutamide); Arm D (EBRT, STAD, apalutamide, RT)
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Other: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Procedure: Intensity-Modulated Proton Therapy — Undergo IMPT
  Other Names: IMPT
  Arms: Arm D (EBRT, STAD, apalutamide, RT)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm D (EBRT, STAD, apalutamide, RT)
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Procedure: Magnetic Resonance Imaging — Undergo PET/MR
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MR
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Relugolix — Given PO
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; TAK 385; TAK-385
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm D (EBRT, STAD, apalutamide, RT)
Drug: Triptorelin — Given IM
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY-25650; CL-118,532; Detryptoreline
Radiation: Volume Modulated Arc Therapy — Undergo VMAT
  Other Names: VMAT; Volumetric Modulated Arc Therapy (procedure)
  Arms: Arm D (EBRT, STAD, apalutamide, RT)

SUMMARY:
This phase III trial tests two questions by two separate comparisons of therapies. The first question is whether enhanced therapy (apalutamide in combination with abiraterone + prednisone) added to standard of care (prostate radiation therapy and short term androgen deprivation) is more effective compared to standard of care alone in patients with prostate cancer who experience biochemical recurrence (a rise in the blood level of prostate specific antigen [PSA] after surgical removal of the prostate cancer).

A second question tests treatment in patients with biochemical recurrence who show prostate cancer spreading outside the pelvis (metastasis) by positron emission tomography (PET) imaging. In these patients, the benefit of adding metastasis-directed radiation to enhanced therapy (apalutamide in combination with abiraterone + prednisone) is tested.

Diagnostic procedures, such as PET, may help doctors look for cancer that has spread to the pelvis. Androgens are hormones that may cause the growth of prostate cancer cells. Apalutamide may help fight prostate cancer by blocking the use of androgens by the tumor cells. Metastasis-directed targeted radiation therapy uses high energy rays to kill tumor cells and shrink tumors that have spread. This trial may help doctors determine if using PET results to deliver more tailored treatment (i.e., adding apalutamide, with or without targeted radiation therapy, to standard of care treatment) works better than standard of care treatment alone in patients with biochemical recurrence of prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. For patients without PET-evidence of extrapelvic metastases, to evaluate whether the addition of enhanced systemic therapy to standard of care (SOC) salvage radiation therapy (RT) could prolong progression-free survival (PFS).

II. For patients with PET-evidence of extrapelvic metastases, to evaluate whether the addition of metastasis-directed RT to enhanced systemic therapy and SOC salvage RT could prolong PFS.

III. To compare overall quality of life, measured by Functional Assessment of Cancer Therapy - Prostate (FACT-P) total score, at 6 months between the two sets of treatment arms (A with B and C with D). (QUALITY OF LIFE [QOL] OBJECTIVE)

SECONDARY OBJECTIVES:

I. To evaluate overall survival in each arm. II. To evaluate event-free survival in each arm. III. To evaluate time to prostate-specific antigen (PSA) progression in each arm.

IV. To assess the incidence of adverse events with the addition of enhanced systemic therapy in patients without PET-evidence of extrapelvic metastases.

V. To assess the incidence of adverse events with local ablative metastasis-directed RT for PET-positive metastatic disease in patients with PET-evidence of extrapelvic metastases.

VI. To estimate the detection rate of PET at the patient and regional level, and to evaluate its concordance with the follow-up Food and Drug Administration (FDA)-approved conventional imaging modalities (CIM) (as available) considered standard-of-care per institution, including computed tomography (CT), bone scintigraphy, magnetic resonance imaging (MRI) and PET imaging.

VII. To determine the distribution of PET-positive lesions among anatomic sites (prostate fossa, intrapelvic soft tissue/lymph node, extrapelvic soft tissue/lymph node, and bone metastases) in patients with post-radical prostatectomy (RP) biochemical recurrence (BCR), correlated with PSA (level, doubling time, velocity) and other relevant clinical parameters.

VIII. To compare the change in overall QOL, measured by FACT-P total score, from baseline to 6 months between the two sets of treatment arms (A with B and C with D). (QOL OBJECTIVE) IX. To compare patient-reported fatigue (Functional Assessment of Chronic Illness Therapy [FACIT]-Fatigue scores) at 6 months between the two sets of treatment arms (A with B and C with D). (QOL OBJECTIVE) X. To compare patient-reported overall QOL (FACT-P scores), fatigue (FACIT-Fatigue scores) and pain interference (patient reported outcomes measurement information system [PROMIS] Pain Interference Short Form 4a) between the two sets of treatment arms (A with B and C with D) at the time of disease progression. (QOL OBJECTIVE)

EXPLORATORY OBJECTIVES:

I.To determine the value of repeat PET (PET2) at time of second PSA progression, clinical concern for progression, or 12 months after completion of enhanced systemic therapy, whichever comes first to assess response to therapy (enhanced systemic therapy +/- focal RT and/or androgen deprivation therapy [ADT]) compared to available standard response assessments (PSA and conventional imaging modalities [CIM]).

II. To compare cognitive function, measured by FACT - cognitive function (Cog) peritoneal cancer index (PCI) and total scores, between the three treatment arms receiving enhanced systemic treatment with ADT and apalutamide (Arms B, C, and D) and antiandrogen therapy (ADT) alone (Arm A) at 6 and 12 month. (QOL OBJECTIVE) III. To compare the change in cognitive function, measured by change in FACT-Cog PCI and total scores, from baseline to 6 and baseline to 12 months, between the three treatment arms receiving enhanced systemic treatment with ADT and apalutamide (Arms B, C, and D) and ADT alone (Arm A) at 6 and 12 months. (QOL OBJECTIVE) IV. To characterize longitudinal change in cognitive function between baseline and 24 months in patients with prostate cancer receiving treatment for biochemical recurrence (BCR) and define clinical and disease related characteristics associated with greater cognitive change by the FACT-Cog PCI and total scores. (QOL OBJECTIVE)

OUTLINE:

STEP 0: Patients undergo SOC PET/CT or PET/MR scan at baseline. Patients randomized to Arms C or D and receiving fluciclovine F18 intravenously (IV) undergo a repeat PET2 at time of PSA progression or clinical concerns for progression or 12 months after completion of enhanced systemic therapy, whichever occurs first. Patients in Arm C or D using another tracer for PET1 do not undergo PET2.

STEP 1: Patients are randomized to 1 of 4 arms based on results of fluciclovine F18 PET/CT or PET/MR in Step 0.

ARM A (PET NEGATIVE FOR EXTRA PELVIC-METASTASES): Patients undergo SOC external beam radiation therapy (EBRT) for 6 months. Patients also receive goserelin acetate subcutaneously (SC), leuprolide acetate intramuscularly (IM), triptorelin IM, relugolix orally (PO), or degarelix SC for 6 months starting up to 3 months prior to EBRT but no later than 7 days after start of EBRT. All treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.

ARM B (PET NEGATIVE FOR EXTRA PELVIC-METASTASES): Patients undergo SOC EBRT and receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC as in Arm A. Patients also receive apalutamide PO once daily (QD) for 6 months in the absence of disease progression or unacceptable toxicity.

ARM C: (PET POSITIVE FOR EXTRA PELVIC-METASTASES): Patients undergo SOC EBRT and receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC as in Arm A. Patients also receive apalutamide PO QD as in Arm B.

ARM D (PET POSITIVE FOR EXTRA PELVIC-METASTASES): Patients undergo SOC EBRT and receive goserelin acetate SC, leuprolide acetate IM, triptorelin IM, relugolix PO, or degarelix SC as in Arm A and apalutamide PO QD as in Arm B. Patients also undergo stereotactic body radiation therapy (SBRT) or 3-dimensional (3D) conformal radiation therapy (CRT), intensity-modulated radiation therapy (IMRT) (including volume modulated arc therapy [VMAT]), and intensity-modulated proton therapy (IMPT) over 3-10 fractions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for the first 2 years, every 6 months for years 3-5, and then annually for years 6-10.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0: REGISTRATION ELIGIBILITY CRITERIA
* Patient must be male and >= 18 years of age.
* Patient must have had a radical prostatectomy (RP) as definitive therapy for histopathologically-proven prostatic adenocarcinoma
* Patient must have biochemical recurrence (BCR) after RP, defined as follows:

  * If time to BCR, defined as time to first detectable PSA ( > lower limit of normal for assay used) after RP, is < 12 months, a minimum PSA level of >= 0.2 ng/mL and a confirmatory reading of >= 0.2 ng/mL is required, per the American Urological Association (AUA) definition (Note: patients with a persistent PSA reading of at least 0.2 ng/mL are eligible)
  * If time to BCR, defined as time to first detectable PSA (> lower limit of normal for assay used) after RP, is >= 12 months, a minimum absolute PSA of 0.5 ng/mL is required
  * If the patient has a detectable PSA (> lower limit of normal for assay used) at any time after RP AND has an eligible baseline SOC PET (PET1) with at least one positive lesion in any location, then there is no minimum PSA requirement
* Patients must have no definite evidence for extrapelvic metastatic disease by conventional imaging modalities (CIM) (CT abdomen/pelvis or MRI abdomen/pelvis AND bone scintigraphy, or equivalent), within 26 weeks prior to Step 0 registration. If a patient only has a study-eligible PET/CT or PET/MR (i.e., PET done without prior CIM): if the PET is negative for extrapelvic lesions, then baseline CIM is NOT required. If the PET positive for extrapelvic lesions, then patient should have a baseline CT/MRI for soft tissue lesions and/or a bone scan for osseous lesions

  * Study eligible = PET using FDA-approved radiotracer and performed within 16 weeks prior to study registration
* Extra-pelvic metastases is defined as any osseous metastases and/or any extrapelvic soft tissue, lymph nodes and organ metastases; extra-pelvic is defined as superior to common iliac bifurcation, outside of standard prostate bed + whole pelvis nodal RT fields. Baseline PET/CT or PET/MR scan (PET1) is eligible for this study if the SOC PET scan is completed with an FDA approved radiotracer for prostate cancer after Step 0 registration and prior to Step 1 randomization OR up to 16 weeks prior to Step 0 registration
* Patient must be a candidate for SOC post-prostatectomy radiation therapy (RT) to the prostate bed and pelvic nodes with androgen deprivation therapy (ADT)
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient must not have started ADT for biochemical recurrence prior to baseline PET (PET1) imaging. A short course of low-dose anti-androgen such as bicalutamide, given after baseline study PET/CT but prior to study registration, is permitted as a brief temporizing measure in advance of starting protocol-approved SOC ADT.
* Patient must not be enrolled in another therapeutic clinical trial
* Patient must be able to lie flat and still for approximately 20-30 minutes or otherwise tolerate a PET scan and radiation treatment planning and delivery
* Patients undergoing a PET/MR must meet local institutional safety guidelines for MRI
* Patient must not have history of seizures or known condition that may cause predisposal to seizures (e.g., stroke or head trauma resulting in loss of consciousness) within 1 year prior to registration
* Patient must not have history of inflammatory bowel disease or any gastrointestinal disorder affecting absorption that is expected to increase risk of complication from radiotherapy
* Hemoglobin (Hgb) >= 9.0 g/dL (independent of transfusion and/or growth factors within 3 months prior to Step 0 registration) (obtained within 8 weeks prior to Step 0 registration)
* Leukocytes >= 3,000/mcL (obtained within 8 weeks prior to Step 0 registration)
* Absolute neutrophil count >= 1,500/mcL (obtained within 8 weeks prior to Step 0 registration)
* Platelets >= 100,000/mcL (obtained within 8 weeks prior to Step 0 registration)
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (patients with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, must have a direct bilirubin of < 1.5 x ULN to be eligible) (obtained within 8 weeks prior to Step 0 registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (obtained within 8 weeks prior to Step 0 registration)
* Creatine < 1.5 x instituional ULN (or measured creatinine clearance > 30 mL/min)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class I or II (by patient symptoms) or A or B (by objective assessment)
* Patient must not have completed a course of prior pelvic radiation therapy for any reason
* Patient must agree not to father children while on study
* Patient must be English or Spanish speaking to be eligible for the QOL component of the study

  * NOTE: Sites cannot translate the associated QOL forms
* STEP 1: RANDOMIZATION ELIGIBILITY CRITERIA
* Patient must have completed a baseline SOC PET/CT or PET/MR (PET1 scan) using FDA approved radiotracer with results of extra-pelvic metastases involvement known (positive or negative). The PET1 must have been completed after Step 0 registration and prior to Step 1 randomization OR up to 12 weeks prior to Step 0 registration
* For patients with negative extra-pelvic metastases, PET-imaging status of intra-pelvic nodes must be known (positive or negative)
* For patients with positive extra-pelvic metastases (defined as any PET positive lesions outside of standard salvage RT fields [prostate bed +/- typical whole pelvis]), the number of extra-pelvic lesions must be known (1 - 5 or > 5 extra-pelvic lesions)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to radiographic progression by conventional imaging or positron emission tomography (PET), symptomatic disease or death, whichever occurs first, assessed up to 10 years
  The power of the PFS analysis is 85% using one-sided 0.025 level stratified logrank test. The overall type I error will be controlled using an O'Brien-Fleming boundary function
PFS prolongation in patients without PET-evidence of extrapelvic metastases | Up to 10 years
  Will evaluate whether the addition of enhanced systemic therapy to standard of care salvage therapy could prolong PFS in this patient population. Will be an intention-to-treat analysis of all randomized patients and performed in parallel with patients with PET-evidence of extrapelvic metastases.
PFS prolongation in patients with PET-evidence of extrapelvic metastases | Up to 10 years
  Will evaluate whether the addition of metastasis-directed radiation therapy to standard of care salvage therapy and enhanced systemic therapy could prolong PFS in this patient population. Will be an intention-to-treat analysis of all randomized patients and performed in parallel without patients with PET-evidence of extrapelvic metastases.
Quality of life (QOL) | Up to 24 months
  Descriptive statistics will be used to characterize QOL over time in each arm.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death or date last known alive, assessed up to 10 years
  Will be characterized by the method of Kaplan and Meier and a logrank test will be used to compare OS between the two arms in each cohort.
Event-free survival | From randomization to radiographic progression by conventional imaging or PET, symptomatic disease, or initiation of new treatment for the disease or death, whichever occurs first, assessed up to 10 years
  Will be characterized by the method of Kaplan and Meier and a logrank test will be used to compare EFS between the two arms in each cohort.
Time to prostate-specific antigen (PSA) progression | From randomization to documented PSA progression or radiographic progression, whichever occurs first, assessed up to 10 years
  Patients without any progression will be censored at the date of last disease assessment that shows free of PSA progression. Will be characterized by the method of Kaplan and Meier and a logrank test will be used to compare time to PSA progression between the two arms in each cohort.
Incidence of adverse events | Up to 10 years
  Toxicity will be defined using the Common Terminology Criteria for Adverse Events.
Detection rate of fluciclovine F18 (18F-fluciclovine) PET | At time of PSA recurrence, as clinically indicated or 12 months after completion of enhanced systemic therapy (whichever occurs first), assessed up to 10 years
  For the detection rate, the proportion of baseline standard of care 18F-fluciclovine PET (PET1) positive results at the patient and regional (prostate fossa, intrapelvic soft tissue/lymph node, extrapelvic soft tissue/lymph node, and bone metastases) level will be calculated and its 95% confidence interval will be estimated using the Exact method based on the binomial distribution.
Concordance of detection rate with the follow-up conventional imaging modalities (CIM) | At time of PSA recurrence, as clinically indicated or 12 months after completion of enhanced systemic therapy (whichever occurs first), assessed up to 10 years
  Will use Cohen's Kappa coefficient to measure the agreement between dichotomized PET results and the dichotomized CIM results. Baseline CIM comparison will not be performed because as per our study eligibility criteria, baseline CIM will be negative for metastases.
Distribution of 18F-fluciclovine PET-positive lesions among anatomic sites | Baseline
  The rate of 18F-fluciclovine PET-positive lesions will be reported for each anatomic site, including prostate fossa, intrapelvic soft tissue/lymph node, extrapelvic soft tissue/lymph node, and bone metastases. Their confidence intervals will be estimated using the Exact method for the binomial distribution. To evaluate if PSA (level, doubling time, velocity) and other relevant clinical parameters affects the positivity distribution, will use the logistic regression to model with the binary outcome (positive vs. negative from PET) and covariates will include anatomic site, PSA, and other clinical parameters. Will test the interactions between anatomic site and PSA (plus other clinical parameters) to see if the positivity distribution across anatomic site may change according to the levels of the interacted terms. Will use the technique of generalized estimating equation to account for the outcome correlations within subjects.
Value of repeat PET to assess response to therapy compared to standard response assessments | At time of second PSA recurrence or 12 months after completion of enhanced systemic therapy (whichever occurs first), assessed up to 10 years
  Analyses will be conducted to evaluate qualitative visual evidence of 18F-fluciclovine PET positive metastatic lesions and quantitative PET standardized-uptake value (SUV) changes on a lesion-to-lesion basis from 18F-fluciclovine PET1 (baseline) to PET2 on visually determined sites of recurrence and metastatic disease. This will be compared to reference standard-of-care conventional imaging (Prostate Cancer Working Group 2 criteria) and PSA response at PET2 time point to determine PET2 response to therapy. PET2 visual and quantitative assessment will also be compared to PFS in the time-to-event analysis using a log-rank test (PET2 visual assessment) and a Cox proportional hazards regression (PET2 quantitative assessment). PET SUV parameters to be obtained at PET1 and PET2 will include SUVmax, SUVpeak. PET SUV change from PET1 to PET2 will include absolute SUVmax and SUVpeak change (PET2-PET1) and percent change of SUVmax and SUVpeak (% change = 100*[(PET2-PET1)/PET1]).)
Comparison - Functional Assessment of Cancer Therapy (FACT)- prostate (P) | At baseline and 3, 6, 9, 12 months
  For the PET-negative cohort, with 216 analyzable patients in each arm, the study will have about 84% power to detect a 6-point (0.29 standard deviation) difference between the two arms using a two-sample t test with two-sided type I error of 0.05. The power will be greater than 99% if the difference between the two arms is 10 points (0.48 standard deviation). For the PET-positive cohort, with 146 analyzable patients in each arm, the study will have 68% and 98% power to detect a 6-point (0.29 standard deviation) and a 10-point (0.48 standard deviation) differences between the two arms, respectively, using the same test.
Change in FACT-P and Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue | Baseline up to 6 months
  A paired t test will be used to compare FACT-P scores at these two time points in each arm. A two-sample t test will be performed to compare the changes in FACT-P scores from baseline to 6 months between the two arms of each cohort. The FACIT-Fatigue scores at 6 months will be compared between the two arms of each cohort using a two-sample t test.
QOL Assessments at Progression | Up to 10 years
  A paired t test will be used to compare FACT-P total scores, FACIT-Fatigue scores and pain scores at these two time points in each arm. The changes in these scores from baseline to progression will be evaluated in each arm.
FACT- cognitive functioning (Cog) | Up to 12 months
  Will be compared between two groups of patients on this study, patients receiving antiandrogen therapy (ADT) + apalutamide (Arms B, C and D) and patients receiving ADT alone (Arm A), at different time points. To ensure similarity of the three arms with systemic treatments (Arms B, C and D), a comparison in FACT-Cog total scores among these three arms will be performed using the Kruskal-Wallis test before combining them together to be compared with Arm A.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Vapiwala, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (303):
- United States (303):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Tarrant County Hospital District/JPS Health Network, Fort Worth, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming